CLINICAL TRIAL: NCT05277805
Title: The Development and Validation of EMPOWER-UP: a Generic Questionnaire for Measuring Empowerment in Patient-provider Relationships
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: King's College London (Other); Deakin University (Other)
Responsible Party: Principal Investigator, Emilie Haarslev Schröder Marqvorsen, Ph.d. student, MSc, Rigshospitalet, Denmark
Other Study IDs: P-2020-706
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Cancer; Diabetes; Mental Disorder
MeSH Terms: conditions — Neoplasms; Diabetes Mellitus; Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EMPOWER-UP participants: People with cancer, diabetes, or mental disorders answering the EMPOWER-UP questionnaire
  Interventions: Other: EMPOWER-UP questionnaire

INTERVENTIONS:
Other: EMPOWER-UP questionnaire — Participants are asked to respond to the EMPOWER-UP questionnaire to test the psychometric properties of the questionnaire.

SUMMARY:
Empowerment is widely acknowledged as an important approach in long-term care. The concept relates to the individual's ability to manage their own life and make rational decisions. Despite good intentions of working empowerment-based, research has shown that it can be difficult to realize and achieve in everyday practice within the healthcare system. To this date, no measurement instrument (questionnaire) exists that evaluate people's perceptions of whether their relationship with a healthcare provider promotes their empowerment process. The EMPOWER-UP questionnaire was therefore developed to provide such a measure. The EMPOWER-UP study aims to finalize the development process of the questionnaire and to test whether it is a valid and reliable measure.

People at the age of 18 years or above can participate if they have ever been diagnosed with a type of cancer, diabetes, or a mental illness and because of that diagnosis have been in contact with the healthcare system within the past six months.

The study is conducted online and requires participants to fill out an online questionnaire on a single occasion. Participation is expected to take no more than 10-15 minutes.

By participating, people may experience an increased awareness as to the nature of their interactions with healthcare providers. For some, this awareness may be beneficial and may alone enable them to ask for better care, while others may experience it as a burden if they are not able to seek better care.

By participating, people are helping to ensure that EMPOWER-UP will be a good questionnaire that may help raise awareness of the quality of relationships within the healthcare system and in term lead to better care.

The study is led by a team of researchers at the Danish University Hospital Rigshospitalet and the University of Copenhagen, Denmark.

The UK lead of the study is located at King's College London, UK. The Australian lead of the study is located at Deakin University, Melbourne, Australia.

This study is financially supported by the Novo Nordisk Foundation's Steno Collaborative Grant and by the Trygfonden foundation (Denmark)

ELIGIBILITY:
Inclusion Criteria:

* Ever diagnosed with cancer, diabetes, or a mental disorder AND have had an interaction with a healthcare provider concerning their cancer/diabetes/mental disorder diagnosis within the past six months (relating to e.g. treatment or follow-up consultations)

Exclusion Criteria:

* Unable to read and understand Danish (for danish participants) or English (for UK and australian participants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People are invited to participate through patient organizations, disease-specific patient boards, general care clinics, and outpatient clinics at hospitals in Denmark, the UK, and Australia
Sampling Method: Non-Probability Sample
Enrollment: 526 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2023-08-23 (Estimated)

PRIMARY OUTCOMES:
Relational empowerment | Baseline
  EMPOWER-UP questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Zoffmann, Professor, Study Chair — Rigshospitalet, Denmark
Locations (3):
- Deakin University, Online, Melbourne, Australia
- Rigshospitalet, online, Copenhagen, Denmark
- King's College London, online, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Danish data collection URL — https://redcap.link/EMPOWER-UP-da
- See also: UK data collection URL — https://redcap.link/EMPOWER-UP-EN
- See also: Australian data collection — https://redcap.link/EMPOWER-UP-aus